CLINICAL TRIAL: NCT00455533
Title: A Randomized Phase II Biomarker Neoadjuvant Study of Sequential AC Followed by Ixabepilone Compared to Sequential AC Followed by Paclitaxel in Women With Early Stage Breast Cancer
Brief Title: Study to Assess Effectiveness of Giving Combination of Standard Chemotherapy Drugs Versus Combination of Standard Chemotherapy and New Drug Ixabepilone When Given Before Surgical Removal of Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-100; EUDRACT 2006-003047-24
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Results first posted 2011-04-04 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Epothilones; Paclitaxel; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Ixabepilone; Drug: Cyclophosphamide; Drug: Doxorubicin
- B (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Cyclophosphamide; Drug: Doxorubicin

INTERVENTIONS:
Drug: Ixabepilone — Intravenous Solution, intravenous (IV), 40mg/m², Day 1 every 21 days, 12 Weeks
  Other Names: Epothilone; IXEMPRA®; BMS-247550
  Arms: A
Drug: Paclitaxel — Intravenous Solution, IV, 80mg/m², Weekly, 12 Weeks
  Arms: B
Drug: Cyclophosphamide — Intravenous Solution, IV, 600mg/m², Day 1 every 21 days, 12 Weeks
Drug: Doxorubicin — Intravenous Solution, IV, 60mg/m², Day 1 every 21 days, 12 Weeks

SUMMARY:
The study will evaluate the effectiveness of ixabepilone when given after doxorubicin plus cyclophosphamide (AC) compared to standard treatment of paclitaxel given after doxorubicin plus cyclophosphamide in patients with early stage breast cancer. In addition the study will verify predefined biomarkers as well as discover new biomarkers that could identify patients who are more likely to respond to ixabepilone than standard paclitaxel based therapy.

ELIGIBILITY:
Inclusion criteria

* Histologically confirmed primary invasive adenocarcinoma of the breast , T2-3, N0-3, M0, with tumor size of ≥ 2 cm
* All patients with early stage breast adenocarcinoma may enroll irrespective of receptor status
* No prior treatment for breast cancer excluding therapy for DCIS
* Karnofsky performance status of 80 - 100
* left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram or multiple gated acquisition (MUGA)
* Adequate hematologic, hepatic and renal function

Exclusion Criteria

* women of child-bearing potential (WOCBP) unwilling or unable to use an acceptable method to avoid pregnancy during and up to 8 weeks after the last dose of the investigational drug
* Women who are pregnant or breastfeeding
* Inflammatory or metastatic breast cancer
* Unfit for breast and/or axillary surgery
* Evidence of baseline sensory or motor neuropathy
* Significant history of cardiovascular disease, serious intercurrent illness or infections including known human immu immunodeficiency virus (HIV) infection
* History of prior anthracycline therapy Allergies to any study medication or Cremophor® EL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- United States (10):
  - Comprehensive Cancer Center, Palm Springs, California
  - Northwest Oncology & Hematology Associates, Coral Spring, Florida
  - Florida Cancer Research Institute, Davie, Florida
  - Medical Specialists Of Palm Beaches, Lake Worth, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University Medical Center, Inc, Louisville, Kentucky
  - University Of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albert Einstein Cancer Center, The Bronx, New York
  - Virginia Mason Medical Center, Seattle, Washington
  - Providence Cancer Center, Spokane, Washington
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
- Austria (2):
  - Local Institution, Salzburg
  - Local Institution, Vienna
- France (2):
  - Local Institution, Bordeaux
  - Local Institution, Saint-Herblain
- Germany (3):
  - Local Institution, Düsseldorf
  - Local Institution, Erlangen
  - Local Institution, Jena
- India (8):
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Trivandrum, Kerala
  - Local Institution, Pune, Maharashtra
  - Local Institution, New Delhi, National Capital Territory of Delhi
  - Local Institution, Bhopal
  - Local Institution, Hyderabad
  - Local Institution, Mumbai
  - Local Institution, Vellore
- Local Institution, Bologna, Italy
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Callao, Provincia Constitucional del Callao
- Philippines (3):
  - Local Institution, Cebu City
  - Local Institution, Davao City
  - Local Institution, Quezon City
- Russia (3):
  - Local Institution, Kazan'
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- Local Institution, Seoul, South Korea
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Jaén
  - Local Institution, Lleida
- Local Institution, Taipei, Taiwan
- United Kingdom (2):
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Coventry, Warwickshire

REFERENCES:
- [Derived] Abdel-Fatah TMA, Agarwal D, Liu DX, Russell R, Rueda OM, Liu K, Xu B, Moseley PM, Green AR, Pockley AG, Rees RC, Caldas C, Ellis IO, Ball GR, Chan SYT. SPAG5 as a prognostic biomarker and chemotherapy sensitivity predictor in breast cancer: a retrospective, integrated genomic, transcriptomic, and protein analysis. Lancet Oncol. 2016 Jul;17(7):1004-1018. doi: 10.1016/S1470-2045(16)00174-1. Epub 2016 Jun 14. PMID 27312051
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 384 participants were enrolled in this study; 71 did not receive any study medication.
Groups:
- Doxorubicin / Cyclophosphamide (AC): 60 mg/m^2 doxorubicin and 600 mg/m^2 cyclophosphamide (AC) every 3 weeks for 4 cycles (12 weeks).
- Ixabepilone: ixabepilone 40 mg/m^2 administered intravenously (IV) over 3 hours, every 3 weeks for 4 cycles (12 weeks)
- Paclitaxel: Paclitaxel 80 mg/m^2 administered IV every week for 12 weeks
Period: Period One: Initial Chemotherapy
Arm/Group | Doxorubicin / Cyclophosphamide (AC) | Ixabepilone | Paclitaxel
Started | 313 | 0 | 0
Completed | 295 | 0 | 0
Not Completed | 18 | 0 | 0
Not completed — Adverse Event Not Related to Study Drug | 1 | 0 | 0
Not completed — Disease Progression | 5 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Not Reported | 1 | 0 | 0
Not completed — Other--Need Reasons | 2 | 0 | 0
Not completed — Study Drug Toxicity | 2 | 0 | 0
Not completed — Subject Request to Discontinue Study | 1 | 0 | 0
Not completed — Subject No Longer Meets Study Criteria | 2 | 0 | 0
Not completed — Subject Withdrew Consent | 2 | 0 | 0
Period: Period Two: Randomized Period
Arm/Group | Doxorubicin / Cyclophosphamide (AC) | Ixabepilone | Paclitaxel
Started | 0 | 145 (148 randomized, 145 randomized and treated with ixabepilone) | 144 (147 randomized, 144 randomized and treated with paclitaxel)
Completed | 0 | 139 | 138
Not Completed | 0 | 6 | 6
Not completed — Death | 0 | 0 | 3
Not completed — Disease Progression | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other - need reasons | 0 | 1 | 0
Not completed — Study Drug Toxicity | 0 | 2 | 0
Not completed — Subject Withdrew Consent | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone (Randomized Population): ixabepilone 40 mg/m^2 administered intravenously (IV) over 3 hours, every 3 weeks for 4 cycles (12 weeks)
- Paclitaxel (Randomized Population): paclitaxel 80 mg/m^2 administered IV every week for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Ixabepilone (Randomized Population) | Paclitaxel (Randomized Population) | Total
Number analyzed (Participants) | 148 | 147 | 295
Age, Continuous [Median (Full Range); unit: years] | 48.0 [25.0 to 79.0] | 46.0 [26.0 to 74.0] | 48.0 [25.0 to 79.0]
Age, Customized [Number; unit: participants]
  <65 years | 134 | 137 | 271
  >=65 years | 14 | 10 | 24
  <50 years | 85 | 82 | 167
  >=50 years | 63 | 65 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 147 | 295
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 74 | 76 | 150
  Black/African American | 7 | 4 | 11
  Asian Indian | 22 | 28 | 50
  Chinese | 16 | 12 | 28
  Asian Other | 17 | 14 | 31
  Unknown or Not Reported | 12 | 13 | 25
Karnofsky Performance Status-Baseline [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0-100, the lower the score, the worse the survival for most serious illnesses.
  participants
    100 - Normal no complaints; no evidence of disease | 107 | 103 | 210
    90 - Normal activity; minor signs of disease | 28 | 39 | 67
    80 - Activity with effort; some signs of disease | 13 | 5 | 18
    70 - Unable to carry on normal activity | 0 | 0 | 0
    <=60 Needs increasing assistance up to Death (0) | 0 | 0 | 0
Menopausal Status [Number; unit: Participants]
  Pre-Menopausal | 71 | 75 | 146
  Peri-Menopausal | 6 | 6 | 12
  Post-Menopausal | 67 | 64 | 131
  Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Pathologic Complete Response (pCR)
Description: The pCR was defined as no histologic evidence of residual invasive adenocarcinoma in the breast and axillary lymph nodes, with or without the presence of ductal carcinoma in situ (DCIS) in the breast.
Time Frame: at surgery (performed 4-6 weeks after the last dose of 12 weeks of therapy)
Population: All randomized participants
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 148 | 147
Percentage of Participants | 24.3 [18.6 to 30.8] | 25.2 [19.4 to 31.7]
Statistical Analysis 1: Comparison: Ixabepilone vs Paclitaxel; Test type: Superiority or Other; p = 0.8921, Fisher Exact
Statistical Analysis 2: Comparison: Ixabepilone vs Paclitaxel; Test type: Superiority or Other; p = 0.8966, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 90% CI 2-sided [0.60 to 1.55]
Statistical Analysis 3: Comparison: Ixabepilone vs Paclitaxel; Test type: Superiority or Other; difference in pCR = -0.6, 95% CI 2-sided [-7.9 to 6.7] — The difference in pCR rates and the confidence interval computed using the method of DerSimonian and Laird stratified by tumor size at baseline, estrogen receptor status, and clinical response to AC

2. Secondary Outcome: Percentage of Participants Achieving Clinical Objective Response
Description: Clinical response was defined as the number of participants who achieved modified World Health Organization's tumor response criteria of clinical complete response (complete disappearance of all clinically palpable detectable malignant disease and/or disappearance of radiological evidence of tumor in the breast and ipsilateral axillary lymph nodes) or clinical partial response (clinical evidence of a reduction in total tumor size of >= 50% in the overall sum of the products of diameters of breast and axillary lesions), divided by the number of randomized participants in that arm.
Time Frame: after the last dose of either ixabepilone or paclitaxel (at 12 weeks) but before surgery (4-6 weeks after the last dose of 12 weeks of therapy)
Population: All randomized participants
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 148 | 147
Percentage of Participants | 81.1 [75.0 to 86.2] | 77.6 [71.2 to 83.1]

3. Secondary Outcome: Percentage of Participants Requiring Breast Conservation Surgery
Description: Number of randomized participants requiring breast conservation surgery following study treatment.
Time Frame: at surgery (performed 4-6 weeks after the last dose of 12 weeks of therapy)
Population: All randomized participants
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 148 | 147
Percentage of Participants | 41.9 [35.1 to 49.0] | 32.7 [26.3 to 39.6]

4. Secondary Outcome: Percentage of Participants Achieving Combined pCR and Minimal Residual Cancer Burden (RCB) 1
Description: Combined pCR and RCB-1 was defined as participants with no histologic evidence of residual invasive adenocarcinoma in the breast and axillary lymph nodes, with or without the presence of DCIS in the breast plus subjects with RCB-1 following the RCB calculation based on data entered by the investigator sites in each arm.
Time Frame: at surgery (performed 4-6 weeks after the last dose of 12 weeks of therapy)
Population: All randomized participants
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 148 | 147
Percentage of Participants | 30.4 [24.2 to 37.2] | 33.3 [26.9 to 40.3]
Statistical Analysis 1: Comparison: Ixabepilone vs Paclitaxel; Test type: Superiority or Other; p = 0.6186, Fisher Exact
Statistical Analysis 2: Comparison: Ixabepilone vs Paclitaxel; Test type: Superiority or Other; p = 0.5806, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.86, 90% CI 2-sided [0.56 to 1.34]
Statistical Analysis 3: Comparison: Ixabepilone vs Paclitaxel; Test type: Superiority or Other; difference = -2.5, 90% CI 2-sided [-11 to 6.0] — The difference in pCR/RCB-I rates and the confidence interval computed using the method of DerSimonian and Laird stratified by tumor size at baseline, estrogen receptor status, and clinical response to AC

5. Secondary Outcome: Randomized Participants With Non-missing pCR & Biomarker Expression (GENE [Probe Set]), to Explore Whether Gene Expression Patterns for GTSE1, Isoforms of β-tubulin, Kallikreins 5, 6, 10 Are Differentially Predictive of pCR
Description: Relevance of biomarker in differentiation between ixabepilone & paclitaxel evaluated by logistic regression with pCR as response. Statistical analyses include: 1) the likelihood ratio test between the full model (PCR~Biomarker:Treatment:estrogen receptor [ER]) & reduced model (PCR~Treatment:ER); 2) the likelihood ratio test between the full model (PCR~Biomarker:Treatment) & reduced model (PCR~Biomarker+Treatment); 3) the contrast of the interaction between treatment & biomarker expression within ER Negative subjects from the full model(PCR~Biomarker:Treatment:ER). A:B represents A,B & A*B.
Time Frame: pCR evaluated at time of surgery (performed 4-6 weeks after the last dose of 12 weeks of therapy); mandatory tumor tissue biopsy obtained prior to treatment.
Measure: Number; unit: participants
Arm/Group | Randomized Participants
Number analyzed (Participants) | 295
participants
  ABCB1 (209993_at) | 245
  ABCB1 /// ABCB4 (209994_s_at) | 245
  BRCA1 (211851_x_at) | 245
  BRCA1 (204531_s_at) | 245
  ERCC1 (203719_at) | 245
  ERCC1 (203720_s_at) | 245
  GTSE1 (204315_s_at) | 245
  GTSE1 (204317_at) | 245
  GTSE1 (215942_s_at) | 245
  GTSE1 (204318_s_at) | 245
  GTSE1 (211040_x_at) | 245
  KLK10 (209792_s_at) | 245
  KLK10 (215808_at) | 245
  KLK5 (222242_s_at) | 245
  KLK6 (204733_at) | 245
  RRM1 (201476_s_at) | 245
  RRM1 (201477_s_at) | 245
  TUBB (211714_x_at) | 245
  TUBB (212320_at) | 245
  TUBB (209026_x_at) | 245
  TUBB1 (208601_s_at) | 245
  TUBB2A (204141_at) | 245
  TUBB2A /// TUBB2B (209372_x_at) | 245
  TUBB2B (214023_x_at) | 245
  TUBB2C (208977_x_at) | 245
  TUBB2C (213726_x_at) | 245
  TUBB4 (212664_at) | 245
  TUBB6 (209191_at) | 245
  TYMS (202589_at) | 245
  TYMS (217684_at) | 245
Statistical Analysis 1: Comparison: Randomized Participants; ABCB1 (209993_at); Test type: Superiority or Other; p = 0.4115, Regression, Logistic — P Value 1 is from the likelihood ratio test between the full model: (PCR ~ Biomarker: Treatment: ER) and the reduced model: (PCR ~ Treatment : ER); p-value not adjusted for multiple comparison
Statistical Analysis 2: Comparison: Randomized Participants; ABCB1 209993_at; Test type: Superiority or Other; p = 0.1629, Regression, Logistic — P Value 2 is from the likelihood ratio test between the full model: (PCR ~ Biomarker: Treatment) and the reduced model: (PCR ~ Biomarker + Treatment); p-value not adjusted for multiple comparison
Statistical Analysis 3: Comparison: Randomized Participants; ABCB1 209993_at; Test type: Superiority or Other; p = 0.5074, Regression, Logistic — P Value 3 is the contrast of the interaction between treatment and biomarker expression within ER Negative subjects from the full model:(PCR ~ Biomarker : Treatment : ER); p-value not adjusted for multiple comparison
Statistical Analysis 4: Comparison: Randomized Participants; ABCB1 /// ABCB4 209994_s_at; Test type: Superiority or Other; p = 0.5530, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 5: Comparison: Randomized Participants; ABCB1 /// ABCB4 209994_s_at; Test type: Superiority or Other; p = 0.1845, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 6: Comparison: Randomized Participants; ABCB1 /// ABCB4 209994_s_at; Test type: Superiority or Other; p = 0.3538, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 7: Comparison: Randomized Participants; BRCA1 211851_x_at; Test type: Superiority or Other; p = 0.9751, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 8: Comparison: Randomized Participants; BRCA1 211851_x_at; Test type: Superiority or Other; p = 0.8874, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 9: Comparison: Randomized Participants; BRCA1 211851_x_at; Test type: Superiority or Other; p = 0.6907, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 10: Comparison: Randomized Participants; BRCA1 204531_s_at; Test type: Superiority or Other; p = 0.8052, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 11: Comparison: Randomized Participants; BRCA1 204531_s_at; Test type: Superiority or Other; p = 0.5031, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 12: Comparison: Randomized Participants; BRCA1 204531_s_at; Test type: Superiority or Other; p = 0.7588, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 13: Comparison: Randomized Participants; ERCC1 203719_at; Test type: Superiority or Other; p = 0.1542, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 14: Comparison: Randomized Participants; ERCC1 203719_at; Test type: Superiority or Other; p = 0.0235, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 15: Comparison: Randomized Participants; ERCC1 203719_at; Test type: Superiority or Other; p = 0.3612, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 16: Comparison: Randomized Participants; ERCC1 203720_s_at; Test type: Superiority or Other; p = 0.1840, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 17: Comparison: Randomized Participants; ERCC1 203720_s_at; Test type: Superiority or Other; p = 0.0942, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 18: Comparison: Randomized Participants; ERCC1 203720_s_at; Test type: Superiority or Other; p = 0.5327, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 19: Comparison: Randomized Participants; GTSE1 204315_s_at; Test type: Superiority or Other; p = 0.8847, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 20: Comparison: Randomized Participants; GTSE1 204315_s_at; Test type: Superiority or Other; p = 0.8947, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 21: Comparison: Randomized Participants; GTSE1 204315_s_at; Test type: Superiority or Other; p = 0.4085, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 22: Comparison: Randomized Participants; GTSE1 204317_at; Test type: Superiority or Other; p = 0.1119, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 23: Comparison: Randomized Participants; GTSE1 204317_at; Test type: Superiority or Other; p = 0.0250, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 24: Comparison: Randomized Participants; GTSE1 204317_at; Test type: Superiority or Other; p = 0.3569, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 25: Comparison: Randomized Participants; GTSE1 215942_s_at; Test type: Superiority or Other; p = 0.4103, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 26: Comparison: Randomized Participants; GTSE1 215942_s_at; Test type: Superiority or Other; p = 0.1490, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 27: Comparison: Randomized Participants; GTSE1 215942_s_at; Test type: Superiority or Other; p = 0.5590, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 28: Comparison: Randomized Participants; GTSE1 204318_s_at; Test type: Superiority or Other; p = 0.4796, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 29: Comparison: Randomized Participants; GTSE1 204318_s_at; Test type: Superiority or Other; p = 0.2794, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 30: Comparison: Randomized Participants; GTSE1 204318_s_at; Test type: Superiority or Other; p = 0.1646, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 31: Comparison: Randomized Participants; GTSE1 211040_x_at; Test type: Superiority or Other; p = 0.0782, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 32: Comparison: Randomized Participants; GTSE1 211040_x_at; Test type: Superiority or Other; p = 0.1407, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 33: Comparison: Randomized Participants; GTSE1 211040_x_at; Test type: Superiority or Other; p = 0.2369, Regression, Logistic — P Value 3 is the contrast of the interaction between treatment and biomarker expression within ER Negative subjects from the full model:(PCR ~ Biomarker : Treatment : ER; p-value not adjusted for multiple comparison
Statistical Analysis 34: Comparison: Randomized Participants; KLK10 209792_s_at; Test type: Superiority or Other; p = 0.7756, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 35: Comparison: Randomized Participants; KLK10 209792_s_at; Test type: Superiority or Other; p = 0.2623, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 36: Comparison: Randomized Participants; KLK10 209792_s_at; Test type: Superiority or Other; p = 0.3147, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 37: Comparison: Randomized Participants; KLK10 215808_at; Test type: Superiority or Other; p = 0.2885, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 38: Comparison: Randomized Participants; KLK10 215808_at; Test type: Superiority or Other; p = 0.7187, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 39: Comparison: Randomized Participants; KLK10 215808_at; Test type: Superiority or Other; p = 0.6017, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 40: Comparison: Randomized Participants; KLK5 222242_s_at; Test type: Superiority or Other; p = 0.4500, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 41: Comparison: Randomized Participants; KLK5 222242_s_at; Test type: Superiority or Other; p = 0.0952, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 42: Comparison: Randomized Participants; KLK5 222242_s_at; Test type: Superiority or Other; p = 0.7069, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 43: Comparison: Randomized Participants; KLK6 204733_at; Test type: Superiority or Other; p = 0.4767, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 44: Comparison: Randomized Participants; KLK6 204733_at; Test type: Superiority or Other; p = 0.6191, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 45: Comparison: Randomized Participants; KLK6 204733_at; Test type: Superiority or Other; p = 0.5276, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 46: Comparison: Randomized Participants; RRM1 201476_s_at; Test type: Superiority or Other; p = 0.3323, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 47: Comparison: Randomized Participants; RRM1 201476_s_at; Test type: Superiority or Other; p = 0.1025, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 48: Comparison: Randomized Participants; RRM1 201476_s_at; Test type: Superiority or Other; p = 0.1715, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 49: Comparison: Randomized Participants; RRM1 201477_s_at; Test type: Superiority or Other; p = 0.1070, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 50: Comparison: Randomized Participants; RRM1 201477_s_at; Test type: Superiority or Other; p = 0.2751, Regression, Logistic — P Value 2 is from the likelihood ratio test between the full model: (PCR ~ Biomarker: Treatment) and the reduced model: (PCR ~ Biomarker + Treatment; p-value not adjusted for multiple comparison
Statistical Analysis 51: Comparison: Randomized Participants; RRM1 201477_s_at; Test type: Superiority or Other; p = 0.0276, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 52: Comparison: Randomized Participants; TUBB 211714_x_at; Test type: Superiority or Other; p = 0.1689, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 53: Comparison: Randomized Participants; TUBB 211714_x_at; Test type: Superiority or Other; p = 0.0769, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 54: Comparison: Randomized Participants; TUBB 211714_x_at; Test type: Superiority or Other; p = 0.1058, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 55: Comparison: Randomized Participants; TUBB 212320_at; Test type: Superiority or Other; p = 0.6406, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 56: Comparison: Randomized Participants; TUBB 212320_at; Test type: Superiority or Other; p = 0.1733, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 57: Comparison: Randomized Participants; TUBB 212320_at; Test type: Superiority or Other; p = 0.2631, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 58: Comparison: Randomized Participants; TUBB 209026_x_at; Test type: Superiority or Other; p = 0.2170, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 59: Comparison: Randomized Participants; TUBB 209026_x_at; Test type: Superiority or Other; p = 0.0868, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 60: Comparison: Randomized Participants; TUBB 209026_x_at; Test type: Superiority or Other; p = 0.1117, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 61: Comparison: Randomized Participants; TUBB1 (208601_s_at); Test type: Superiority or Other; p = 0.4943, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 62: Comparison: Randomized Participants; TUBB1 208601_s_at; Test type: Superiority or Other; p = 0.5190, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 63: Comparison: Randomized Participants; TUBB1 208601_s_at; Test type: Superiority or Other; p = 0.7350, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 64: Comparison: Randomized Participants; TUBB2A 204141_at; Test type: Superiority or Other; p = 0.3820, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 65: Comparison: Randomized Participants; TUBB2A 204141_at; Test type: Superiority or Other; p = 0.9290, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 66: Comparison: Randomized Participants; TUBB2A 204141_at; Test type: Superiority or Other; p = 0.0699, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 67: Comparison: Randomized Participants; TUBB2A /// TUBB2B 209372_x_at; Test type: Superiority or Other; p = 0.3515, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 68: Comparison: Randomized Participants; TUBB2A /// TUBB2B 209372_x_at; Test type: Superiority or Other; p = 0.2128, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 69: Comparison: Randomized Participants; TUBB2A /// TUBB2B 209372_x_at; Test type: Superiority or Other; p = 0.1275, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 70: Comparison: Randomized Participants; TUBB2B 214023_x_at; Test type: Superiority or Other; p = 0.2158, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 71: Comparison: Randomized Participants; TUBB2B 214023_x_at; Test type: Superiority or Other; p = 0.0266, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 72: Comparison: Randomized Participants; TUBB2B 214023_x_at; Test type: Superiority or Other; p = 0.3636, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 73: Comparison: Randomized Participants; TUBB2C 208977_x_at; Test type: Superiority or Other; p = 0.9479, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 74: Comparison: Randomized Participants; TUBB2C 208977_x_at; Test type: Superiority or Other; p = 0.3753, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 75: Comparison: Randomized Participants; TUBB2C 208977_x_at; Test type: Superiority or Other; p = 0.5477, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 76: Comparison: Randomized Participants; TUBB2C 213726_x_at; Test type: Superiority or Other; p = 0.4760, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 77: Comparison: Randomized Participants; TUBB2C 213726_x_at; Test type: Superiority or Other; p = 0.3314, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 78: Comparison: Randomized Participants; TUBB2C 213726_x_at; Test type: Superiority or Other; p = 0.1005, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 79: Comparison: Randomized Participants; TUBB4 212664_at; Test type: Superiority or Other; p = 0.1180, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 80: Comparison: Randomized Participants; TUBB4 212664_at; Test type: Superiority or Other; p = 0.1580, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 81: Comparison: Randomized Participants; TUBB4 212664_at; Test type: Superiority or Other; p = 0.4385, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 82: Comparison: Randomized Participants; TUBB6 209191_at; Test type: Superiority or Other; p = 0.7324, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 83: Comparison: Randomized Participants; TUBB6 209191_at; Test type: Superiority or Other; p = 0.2657, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 84: Comparison: Randomized Participants; TUBB6 209191_at; Test type: Superiority or Other; p = 0.5637, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 85: Comparison: Randomized Participants; TYMS 202589_at; Test type: Superiority or Other; p = 0.4473, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 86: Comparison: Randomized Participants; TYMS 202589_at; Test type: Superiority or Other; p = 0.3292, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 87: Comparison: Randomized Participants; TYMS 202589_at; Test type: Superiority or Other; p = 0.2054, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 88: Comparison: Randomized Participants; TYMS 217684_at; Test type: Superiority or Other; p = 0.5226, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 89: Comparison: Randomized Participants; TYMS 217684_at; Test type: Superiority or Other; p = 0.1720, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 90: Comparison: Randomized Participants; TYMS 217684_at; Test type: Superiority or Other; p = 0.3346, Regression, Logistic — [p-value comment as in outcome 5, analysis 3]; p-value not adjusted for multiple comparison

6. Secondary Outcome: Randomized Participants With Non-missing pCR & Biomarker Expression (GENE [Probe Set]) to Explore Whether Gene Expression Patterns for GTSE1, Isoforms of β-tubulin, Kallikreins 5, 6, 10 Are Differentially Predictive of pCR/RCB1
Description: Relevance of biomarker in differentiation between ixabepilone & paclitaxel evaluated by logistic regression with pCR/RCB1 as response. Statistical analyses include: 1) likelihood ratio test between the full model (pCR/RCB1~Biomarker:Treatment: ER) & reduced model (pCR/RCB1~Treatment:ER); 2) likelihood ratio test between the full model (pCR/RCB1 Biomarker:Treatment) & reduced model (pCR/RCB1~Biomarker+Treatment); 3) contrast of the interaction between treatment & biomarker expression within ER Negative subjects from the full model (pCR/RCB1~Biomarker:Treatment:ER). A:B represents A,B & A*B.
Time Frame: pCR evaluated at time of surgery (4-6 weeks after the last dose of therapy); mandatory tumor tissue biopsy obtained prior to treatment.
Measure: Number; unit: participants
Arm/Group | Randomized Participants
Number analyzed (Participants) | 295
participants
  ABCB1 (209993_at) | 245
  ABCB1 /// ABCB4 (209994_s_at) | 245
  BRCA1 (211851_x_at) | 245
  BRCA1 (204531_s_at) | 245
  ERCC1 (203719_at) | 245
  ERCC1 (203720_s_at) | 245
  GTSE1 (204315_s_at) | 245
  GTSE1 (204317_at) | 245
  GTSE1 (215942_s_at) | 245
  GTSE1 (204318_s_at) | 245
  GTSE1 (211040_x_at) | 245
  KLK10 (209792_s_at) | 245
  KLK10 (215808_at) | 245
  KLK5 (222242_s_at) | 245
  KLK6 (204733_at) | 245
  RRM1 (201476_s_at) | 245
  RRM1 (201477_s_at) | 245
  TUBB (211714_x_at) | 245
  TUBB (212320_at) | 245
  TUBB (209026_x_at) | 245
  TUBB1 (208601_s_at) | 245
  TUBB2A (204141_at) | 245
  TUBB2A /// TUBB2B (209372_x_at) | 245
  TUBB2B (214023_x_at) | 245
  TUBB2C (208977_x_at) | 245
  TUBB2C (213726_x_at) | 245
  TUBB4 (212664_at) | 245
  TUBB6 (209191_at) | 245
  TYMS (202589_at) | 245
  TYMS (217684_at) | 245
Statistical Analysis 1: Comparison: Randomized Participants; ABCB1 209993_at; Test type: Superiority or Other; p = 0.5604, Regression, Logistic — P Value 1 is from the likelihood ratio test between the full model: (PCR/RCB1 ~ Biomarker: Treatment: ER) and the reduced model: (PCR/RCB1 ~ Treatment : ER); p-value not adjusted for multiple comparison
Statistical Analysis 2: Comparison: Randomized Participants; ABCB1 209993_at; Test type: Superiority or Other; p = 0.2715, Regression, Logistic — P Value 2 is from the likelihood ratio test between the full model: (PCR/RCB1 ~ Biomarker: Treatment) and the reduced model: (PCR/RCB1 ~ Biomarker + Treatment); p-value not adjusted for multiple comparison
Statistical Analysis 3: Comparison: Randomized Participants; ABCB1 209993_at; Test type: Superiority or Other; p = 0.5268, Regression, Logistic — P Value 3 is the contrast of the interaction between treatment and biomarker expression within ER Negative subjects from the full model:(PCR/RCB1 ~ Biomarker : Treatment : ER); p-value not adjusted for multiple comparison
Statistical Analysis 4: Comparison: Randomized Participants; ABCB1 /// ABCB4 209994_s_at; Test type: Superiority or Other; p = 0.6058, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 5: Comparison: Randomized Participants; ABCB1 /// ABCB4 209994_s_at; Test type: Superiority or Other; p = 0.1918, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 6: Comparison: Randomized Participants; ABCB1 /// ABCB4 209994_s_at; Test type: Superiority or Other; p = 0.6712, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 7: Comparison: Randomized Participants; BRCA1 211851_x_at; Test type: Superiority or Other; p = 0.9195, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 8: Comparison: Randomized Participants; BRCA1 211851_x_at; Test type: Superiority or Other; p = 0.7021, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 9: Comparison: Randomized Participants; BRCA1 211851_x_at; Test type: Superiority or Other; p = 0.3910, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 10: Comparison: Randomized Participants; BRCA1 204531_s_at; Test type: Superiority or Other; p = 0.2909, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 11: Comparison: Randomized Participants; BRCA1 204531_s_at; Test type: Superiority or Other; p = 0.3336, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 12: Comparison: Randomized Participants; BRCA1 204531_s_at; Test type: Superiority or Other; p = 0.2360, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 13: Comparison: Randomized Participants; ERCC1 203719_at; Test type: Superiority or Other; p = 0.0281, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 14: Comparison: Randomized Participants; ERCC1 203719_at; Test type: Superiority or Other; p = 0.0434, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 15: Comparison: Randomized Participants; ERCC1 203719_at; Test type: Superiority or Other; p = 0.0283, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 16: Comparison: Randomized Participants; ERCC1 203720_s_at; Test type: Superiority or Other; p = 0.0151, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 17: Comparison: Randomized Participants; ERCC1 203720_s_at; Test type: Superiority or Other; p = 0.1999, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 18: Comparison: Randomized Participants; ERCC1 203720_s_at; Test type: Superiority or Other; p = 0.0146, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 19: Comparison: Randomized Participants; GTSE1 204315_s_at; Test type: Superiority or Other; p = 0.1185, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 20: Comparison: Randomized Participants; GTSE1 204315_s_at; Test type: Superiority or Other; p = 0.8705, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 21: Comparison: Randomized Participants; GTSE1 204315_s_at; Test type: Superiority or Other; p = 0.0284, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 22: Comparison: Randomized Participants; GTSE1 204317_at; Test type: Superiority or Other; p = 0.0399, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 23: Comparison: Randomized Participants; GTSE1 204317_at; Test type: Superiority or Other; p = 0.0136, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 24: Comparison: Randomized Participants; GTSE1 204317_at; Test type: Superiority or Other; p = 0.0576, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 25: Comparison: Randomized Participants; GTSE1 215942_s_at; Test type: Superiority or Other; p = 0.2245, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 26: Comparison: Randomized Participants; GTSE1 215942_s_at; Test type: Superiority or Other; p = 0.1388, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 27: Comparison: Randomized Participants; GTSE1 215942_s_at; Test type: Superiority or Other; p = 0.0692, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 28: Comparison: Randomized Participants; GTSE1 204318_s_at; Test type: Superiority or Other; p = 0.1058, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 29: Comparison: Randomized Participants; GTSE1 204318_s_at; Test type: Superiority or Other; p = 0.2688, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 30: Comparison: Randomized Participants; GTSE1 204318_s_at; Test type: Superiority or Other; p = 0.0192, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 31: Comparison: Randomized Participants; GTSE1 211040_x_at; Test type: Superiority or Other; p = 0.0033, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 32: Comparison: Randomized Participants; GTSE1 211040_x_at; Test type: Superiority or Other; p = 0.2053, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 33: Comparison: Randomized Participants; GTSE1 211040_x_at; Test type: Superiority or Other; p = 0.0032, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 34: Comparison: Randomized Participants; KLK10 209792_s_at; Test type: Superiority or Other; p = 0.6783, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 35: Comparison: Randomized Participants; KLK10 209792_s_at; Test type: Superiority or Other; p = 0.1630, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 36: Comparison: Randomized Participants; KLK10 209792_s_at; Test type: Superiority or Other; p = 0.2944, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 37: Comparison: Randomized Participants; KLK10 215808_at; Test type: Superiority or Other; p = 0.3727, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 38: Comparison: Randomized Participants; KLK10 215808_at; Test type: Superiority or Other; p = 0.8796, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 39: Comparison: Randomized Participants; KLK10 215808_at; Test type: Superiority or Other; p = 0.8344, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 40: Comparison: Randomized Participants; KLK5 222242_s_at; Test type: Superiority or Other; p = 0.2700, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 41: Comparison: Randomized Participants; KLK5 222242_s_at; Test type: Superiority or Other; p = 0.2624, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 42: Comparison: Randomized Participants; KLK5 222242_s_at; Test type: Superiority or Other; p = 0.0830, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 43: Comparison: Randomized Participants; KLK6 204733_at; Test type: Superiority or Other; p = 0.0849, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 44: Comparison: Randomized Participants; KLK6 204733_at; Test type: Superiority or Other; p = 0.6578, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 45: Comparison: Randomized Participants; KLK6 204733_at; Test type: Superiority or Other; p = 0.0396, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 46: Comparison: Randomized Participants; RRM1 201476_s_at; Test type: Superiority or Other; p = 0.1657, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 47: Comparison: Randomized Participants; RRM1 201476_s_at; Test type: Superiority or Other; p = 0.0675, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 48: Comparison: Randomized Participants; RRM1 201476_s_at; Test type: Superiority or Other; p = 0.1071, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 49: Comparison: Randomized Participants; RRM1 201477_s_at; Test type: Superiority or Other; p = 0.0142, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 50: Comparison: Randomized Participants; RRM1 201477_s_at; Test type: Superiority or Other; p = 0.2465, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 51: Comparison: Randomized Participants; RRM1 201477_s_at; Test type: Superiority or Other; p = 0.0031, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 52: Comparison: Randomized Participants; TUBB 211714_x_at; Test type: Superiority or Other; p = 0.1231, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 53: Comparison: Randomized Participants; TUBB 211714_x_at; Test type: Superiority or Other; p = 0.0849, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 54: Comparison: Randomized Participants; TUBB 211714_x_at; Test type: Superiority or Other; p = 0.2740, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 55: Comparison: Randomized Participants; TUBB 212320_at; Test type: Superiority or Other; p = 0.2383, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 56: Comparison: Randomized Participants; TUBB 212320_at; Test type: Superiority or Other; p = 0.0644, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 57: Comparison: Randomized Participants; TUBB 212320_at; Test type: Superiority or Other; p = 0.2866, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 58: Comparison: Randomized Participants; TUBB 209026_x_at; Test type: Superiority or Other; p = 0.1259, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 59: Comparison: Randomized Participants; TUBB 209026_x_at; Test type: Superiority or Other; p = 0.0718, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 60: Comparison: Randomized Participants; TUBB 209026_x_at; Test type: Superiority or Other; p = 0.3170, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 61: Comparison: Randomized Participants; TUBB1 208601_s_at; Test type: Superiority or Other; p = 0.7844, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 62: Comparison: Randomized Participants; TUBB1 208601_s_at; Test type: Superiority or Other; p = 0.4688, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 63: Comparison: Randomized Participants; TUBB1 208601_s_at; Test type: Superiority or Other; p = 0.8553, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 64: Comparison: Randomized Participants; TUBB2A 204141_at; Test type: Superiority or Other; p = 0.6926, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 65: Comparison: Randomized Participants; TUBB2A 204141_at; Test type: Superiority or Other; p = 0.2222, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 66: Comparison: Randomized Participants; TUBB2A 204141_at; Test type: Superiority or Other; p = 0.4676, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 67: Comparison: Randomized Participants; TUBB2A /// TUBB2B 209372_x_at; Test type: Superiority or Other; p = 0.2036, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 68: Comparison: Randomized Participants; TUBB2A /// TUBB2B 209372_x_at; Test type: Superiority or Other; p = 0.4197, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 69: Comparison: Randomized Participants; TUBB2A /// TUBB2B 209372_x_at; Test type: Superiority or Other; p = 0.0776, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 70: Comparison: Randomized Participants; TUBB2B 214023_x_at; Test type: Superiority or Other; p = 0.4076, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 71: Comparison: Randomized Participants; TUBB2B 214023_x_at; Test type: Superiority or Other; p = 0.0629, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 72: Comparison: Randomized Participants; TUBB2B 214023_x_at; Test type: Superiority or Other; p = 0.2547, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 73: Comparison: Randomized Participants; TUBB2C 208977_x_at; Test type: Superiority or Other; p = 0.7125, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 74: Comparison: Randomized Participants; TUBB2C 208977_x_at; Test type: Superiority or Other; p = 0.6001, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 75: Comparison: Randomized Participants; TUBB2C 208977_x_at; Test type: Superiority or Other; p = 0.5398, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 76: Comparison: Randomized Participants; TUBB2C 213726_x_at; Test type: Superiority or Other; p = 0.3970, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 77: Comparison: Randomized Participants; TUBB2C 213726_x_at; Test type: Superiority or Other; p = 0.5085, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 78: Comparison: Randomized Participants; TUBB2C 213726_x_at; Test type: Superiority or Other; p = 0.1213, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 79: Comparison: Randomized Participants; TUBB4 212664_at; Test type: Superiority or Other; p = 0.0999, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 80: Comparison: Randomized Participants; TUBB4 212664_at; Test type: Superiority or Other; p = 0.1201, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 81: Comparison: Randomized Participants; TUBB4 212664_at; Test type: Superiority or Other; p = 0.1172, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 82: Comparison: Randomized Participants; TUBB6 209191_at; Test type: Superiority or Other; p = 0.6596, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 83: Comparison: Randomized Participants; TUBB6 209191_at; Test type: Superiority or Other; p = 0.3289, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 84: Comparison: Randomized Participants; TUBB6 209191_at; Test type: Superiority or Other; p = 0.3657, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 85: Comparison: Randomized Participants; TYMS 202589_at; Test type: Superiority or Other; p = 0.0275, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 86: Comparison: Randomized Participants; TYMS 202589_at; Test type: Superiority or Other; p = 0.3946, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 87: Comparison: Randomized Participants; TYMS 202589_at; Test type: Superiority or Other; p = 0.0074, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison
Statistical Analysis 88: Comparison: Randomized Participants; TYMS 217684_at; Test type: Superiority or Other; p = 0.2341, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; p-value not adjusted for multiple comparison
Statistical Analysis 89: Comparison: Randomized Participants; TYMS 217684_at; Test type: Superiority or Other; p = 0.0933, Regression, Logistic — [p-value comment as in outcome 6, analysis 2]; p-value not adjusted for multiple comparison
Statistical Analysis 90: Comparison: Randomized Participants; TYMS 217684_at; Test type: Superiority or Other; p = 0.2016, Regression, Logistic — [p-value comment as in outcome 6, analysis 3]; p-value not adjusted for multiple comparison

7. Secondary Outcome: Percentage of Participants With pCR and MDR1 Immunohistochemistry (IHC) Positivity Using Two Pre-Specified Thresholds
Description: Percentage of participants with pCR in MDR1 IHC positive and negative groups using 2 pre-specified thresholds,. The first pre-specified threshold for MDR1-positivity (Mem) =Any membrane staining. The second pre-specified threshold for MDR1-positivity (Mem+Cyto)=Any membrane staining or at least 200 Cytoplasmic H-score.
Time Frame: : pCR evaluated at time of surgery (4-6 weeks after the last dose of 12 weeks of therapy); mandatory tumor tissue biopsy obtained prior to treatment.
Population: Randomized participants with non-missing pCR and biomarker expression
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 111 | 117
percentage of participants
  Mem+Cyto Threshold/Negative Biomarker Status | 0.143 [0.069 to 0.252] | 0.288 [0.193 to 0.4]
  Mem+Cyto Threshold/Positive Biomarker Status | 0.323 [0.225 to 0.433] | 0.259 [0.167 to 0.37]
  Mem Threshold/Negative Biomarker Status | 0.228 [0.158 to 0.312] | 0.284 [0.211 to 0.367]
  Mem Threshold/Negative Biomarker Status | 0.316 [0.147 to 0.53] | 0.2 [0.057 to 0.44]
Statistical Analysis 1: Comparison: Ixabepilone vs Paclitaxel; Mem+Cyto Threshold/Negative Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = -0.145, 90% CI 2-sided [-0.27 to -0.017] — ixabepilone - paclitaxel
Statistical Analysis 2: Comparison: Ixabepilone vs Paclitaxel; Mem+Cyto Threshold/Positive Biomarker STatus; Test type: Superiority or Other; Difference (bootstrap method) = 0.064, 90% CI 2-sided [-0.064 to 0.197] — ixabepilone - paclitaxel
Statistical Analysis 3: Comparison: Ixabepilone vs Paclitaxel; Membrane Threshold/Negative Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = -0.056, 90% CI 2-sided [-0.152 to 0.046] — ixabepilone - paclitaxel
Statistical Analysis 4: Comparison: Ixabepilone vs Paclitaxel; Membrane Threshold/Positive Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = 0.116, 90% CI 2-sided [-0.13 to 0.37] — ixabepilone - paclitaxel

8. Secondary Outcome: Percentage of Participants With pCR/RCB1 and MDR1 Immunohistochemistry (IHC) Positivity Using Two Pre-specified Thresholds
Description: Percentage of participants with pCR/RCB1 in MDR1 IHC positive and negative groups using 2 pre-specified thresholds,. The first pre-specified threshold for MDR1-positivity (Mem) =Any membrane staining. The second pre-specified threshold for MDR1-positivity (Mem+Cyto)=Any membrane staining or at least 200 Cytoplasmic H-score .
Time Frame: pCR evaluated at time of surgery (4-6 weeks after the last dose of 12 weeks of therapy); mandatory tumor tissue biopsy obtained prior to treatment.
Population: Randomized participants with non-missing pCR/RCB1 and biomarker expression
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 111 | 117
percentage of participants
  Mem+Cyto Threshold/Negative Biomarker Status | 0.224 [0.131 to 0.344] | 0.339 [0.237 to 0.453]
  Mem+Cyto Threshold/Positive Biomarker Status | 0.371 [0.268 to 0.483] | 0.362 [0.257 to 0.478]
  Mem Threshold/Negative Biomarker Status | 0.304 [0.226 to 0.393] | 0.363 [0.283 to 0.448]
  Mem Threshold/Negative Biomarker Status | 0.316 [0.147 to 0.53] | 0.267 [0.097 to 0.511]
Statistical Analysis 1: Comparison: Ixabepilone vs Paclitaxel; Mem+Cyto/Negative Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = -0.114, 90% CI 2-sided [-0.258 to 0.22] — ixabepilone - paclitaxel
Statistical Analysis 2: Comparison: Ixabepilone vs Paclitaxel; Mem+Cyto Threshold/Positive Biomarker Status; Test type: Superiority or Other; DIfference (bootstrap method) = 0.009, 90% CI 2-sided [-0.137 to 0.155] — ixabepilone - paclitaxel
Statistical Analysis 3: Comparison: Ixabepilone vs Paclitaxel; Membrane Threshold/Negative Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = -0.058, 90% CI 2-sided [-0.167 to 0.053] — ixabepilone - paclitaxel
Statistical Analysis 4: Comparison: Ixabepilone vs Paclitaxel; Membrane Threshold/Positive Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = 0.049, 90% CI 2-sided [-0.227 to 0.309] — ixabepilone - paclitaxel

9. Secondary Outcome: Percentage of Participants With pCR and MDR1 Immunohistochemistry (IHC) Positivity Using Two Pre-specified Thresholds, Estrogen-Receptor (ER) Negative Participants
Description: Percentage of ER negative participants with pCR and MDR1 immunohistochemistry (IHC) positivity using 2 pre-specified thresholds, stratified by biomarker status. The first pre-specified threshold for MDR1-positivity (Mem)=Any membrane staining. The second pre-specified threshold for MDR1-positivity (Mem+Cyto)=Any membrane staining or at least 200 Cytoplasmic H-score.
Time Frame: as for outcome 8
Population: Randomized estrogen negative participants with non-missing pCR and biomarker expression
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 64 | 70
percentage of participants
  Mem+Cyto Threshold/Negative Biomarker Status | 0.192 [0.079 to 0.363] | 0.483 [0.32 to 0.648]
  Mem+Cyto Threshold/Positive Biomarker Status | 0.447 [0.309 to 0.593] | 0.341 [0.22 to 0.481]
  Mem Threshold/Negative Biomarker Status | 0.327 [0.22 to 0.449] | 0.417 [0.309 to 0.531]
  Mem Threshold/Negative Biomarker Status | 0.417 [0.181 to 0.685] | 0.3 [0.087 to 0.607]
Statistical Analysis 1: Comparison: Ixabepilone vs Paclitaxel; Mem+Cyto Threshold/Negative Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = -0.29, 90% CI 2-sided [-0.482 to -0.094] — ixabepilone - paclitaxel
Statistical Analysis 2: Comparison: Ixabepilone vs Paclitaxel; Mem+Cyto Threshold/Positive Biomarker Status; Test type: Superiority or Other; Difference (boostrap method) = 0.106, 90% CI 2-sided [-0.073 to 0.291] — ixabepilone - paclitaxel
Statistical Analysis 3: Comparison: Ixabepilone vs Paclitaxel; Membrane Threshold/Negative Biomarker Status; Test type: Superiority or Other; Difference (bootstrap method) = -0.09, 90% CI 2-sided [-0.236 to 0.067] — ixabepilone - paclitaxel
Statistical Analysis 4: Comparison: Ixabepilone vs Paclitaxel; Mem+Cyto Threshold/Positive Biomarker Status; Test type: Superiority or Other; Difference (bootsrap method) = 0.117, 90% CI 2-sided [-0.218 to 0.469] — ixabepilone - paclitaxel

10. Secondary Outcome: Prevalence of Biomarker Based on Optimal Threshold (Biomarker Positive Participants)
Description: Percentage of participants having the following optimal biomarker thresholds as computed from the cross-validation method (cutoff of biomarker positive [with 90% confidence interval by Bootstrap method]): Beta 3 Tubulin IHC (45.866 [5, 83.9]); TACC3 mRNA (6.714 [6.312, 7.192]); CAPG mRNA (6.739 [5.728, 7.298]). Optimal thresholds for a 20-gene model and a 26-gene model were also planned; however, these were not determined because preliminary analyses did not indicate that they would not differentiate pCR rates between treatment arm.
Time Frame: pCR evaluated at time of surgery (4-6 weeks after the last dose of 12 weeks of therapy); mandatory tumor tissue biopsy and mRNA samples obtained prior to treatment
Population: Randomized participants with non-missing pCR and biomarker expressions. n=the number of participants with specific biomarker expression.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Randomized Participants: Randomized Participants with non-missing pCR and biomarker expression
Arm/Group | Randomized Participants
Number analyzed (Participants) | 245
Percentage of Participants
  Beta 3 Tubulin IHC (n=231) | 0.394 [0.242 to 0.571]
  Beta 3 Tubulin IHC H-Score (n=231) | 0.299 [0.173 to 0.524]
  Beta 3 Tubulin mRNA (n=245) | 0.392 [0.167 to 0.772]
  TACC3 mRNA (n=245) | 0.514 [0.273 to 0.743]
  CAPG mRNA (n=245) | 0.486 [0.294 to 0.767]

11. Secondary Outcome: Overall Safety Summary: Deaths, Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), Drug-Related AEs, and Most Common Treatment-Related Non-Hematologic Adverse Events (TNAEs) Occuring in >=10% of Participants
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event. By Worst Common Terminology Criteria of Adverse Events (CTCAE Version 3) Grades
Time Frame: prior to the first study treatment, at the beginning of each subsequent cycle, weekly during the treatment period and a minimum of 4 weeks after the last dose of 12 weeks of study therapy
Measure: Number; unit: Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 148 | 147
Participants
  Death | 0 | 2
  Any SAE, Grade (Gr) 1 (mild) | 0 | 0
  Any SAE, Grade 2 (moderate) | 2 | 0
  Any SAE, Grade 3 (severe) | 8 | 6
  Any SAE, Grade 4 (life-threatening) | 6 | 3
  Any SAE, Grade 5 (death) | 0 | 1
  Any SAE, Grade Unknown | 1 | 1
  AE Leading to Discontinuation, Grade 1 (mild) | 0 | 0
  AE Leading to Discontinuation, Grade 2 (moderate) | 3 | 8
  AE Leading to Discontinuation, Grade 3 (severe) | 7 | 4
  AE Leading to Discon, Grade 4 (life-threatening) | 4 | 1
  Any Drug-Related AE, Grade 1 (mild) | 24 | 40
  Any Drug-Related AE, Grade 2 (moderate) | 45 | 54
  Any Drug-Related AE, Grade 3 (severe) | 46 | 24
  Any Drug-Related AE, Grade 4 (life-threatening) | 15 | 3
  TNAE: Peripheral Sensory Neuropathy,Grade 1 (mild) | 36 | 46
  TNAE:Peripheral Sensory Neuropathy,Gr 2 (moderate) | 21 | 21
  TNAE: Peripheral Sensory Neuropathy, Gr 3 (severe) | 6 | 5
  TNAE: Peripheral Sensory Neuropathy, Grade 4 | 0 | 0
  TNAE: Myalgia, Grade 1 (mild) | 18 | 13
  TNAE: Myalgia, Grade 2 (moderate) | 19 | 5
  TNAE: Myalgia, Grade 3 (severe) | 4 | 1
  TNAE: Myalgia, Grade 4 (life-threatening) | 0 | 0
  TNAE: Arthralgia, Grade 1 (mild) | 15 | 12
  TNAE: Arthralgia, Grade 2 (moderate) | 18 | 2
  TNAE: Arthralgia, Grade 3 (severe) | 1 | 0
  TNAE: Arthralgia, Grade 4 (life-threatening) | 0 | 0
  TNAE: Bone Pain, Grade 1 (mild) | 10 | 5
  TNAE: Bone Pain, Grade 2 (moderate) | 11 | 1
  TNAE: Bone Pain, Grade 3 (severe) | 7 | 0
  TNAE: Bone Pain, Grade 4 (life-threatening) | 0 | 0
  TNAE: Fatigue, Grade 1 (mild) | 11 | 12
  TNAE: Fatigue, Grade 2 (moderate) | 11 | 10
  TNAE: Fatigue, Grade 3 (severe) | 5 | 2
  TNAE: Fatigue, Grade 4 (life-threatening) | 0 | 0
  TNAE: Diarrhea, Grade 1 (mild) | 19 | 11
  TNAE: Diarrhea, Grade 2 | 4 | 5
  TNAE: Diarrhea, Grade 3 (severe) | 2 | 2
  TNAE: Diarrhea, Grade 4 (life-threatening) | 0 | 0
  TNAE: Nausea, Grade 1 (mild) | 18 | 16
  TNAE: Nausea, Grade 2 | 6 | 1
  TNAE: Nausea, Grade 3 (severe) | 1 | 0
  TNAE: Nausea, Grade 4 (life-threatening) | 0 | 0
  TNAE: Musculoskeletal Pain, Grade 1 (mild) | 9 | 4
  TNAE: Musculoskeletal Pain, Grade 2 (moderate) | 5 | 1
  TNAE: Musculoskeletal Pain, Grade 3 (severe) | 1 | 1
  TNAE: Musculoskeletal Pain,Gr 4 (life-threatening) | 0 | 0

12. Secondary Outcome: Severity of Any Drug-Related AEs and Gastrointestinal AEs by System Organ Class
Description: MCT=musculoskeletal and connective tissue, GDASC=general disorders and administration site conditions, RTM=respiratory, thoracic and mediastinal disorders, NBMUCP=neoplasms benign, malignant and unspecified (including cysts and polyps). Drug related adverse events are those events with relationship to study therapy of certain, probable, possible or missing. Subjects may have more than one event within a class. Graded by National Cancer Institute Common Terminology Criteria for Adverse Events v3.0. (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death)
Time Frame: as for outcome 11
Population: Ixabepilone- and Paclitaxel-treated participants
Measure: Number; unit: Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 145 | 144
Participants
  Any Drug-Related AEs, Grade (Gr) 1 | 5 | 8
  Any Drug-Related AEs, Gr 2 | 56 | 69
  Any Drug-Related AEs, Gr 3 | 55 | 32
  Any Drug-Related AEs, Gr 4 | 22 | 23
  Any Drug-Related AEs, Gr 5 | 0 | 0
  Gastrointestinal Disorder AEs, Gr 1 | 54 | 52
  Gastrointestinal Disorder AEs, Gr 2 | 42 | 44
  Gastrointestinal Disorder AEs, Gr 3 | 10 | 6
  Gastrointestinal Disorder AEs, Gr 4 | 0 | 0
  Gastrointestinal Disorder AEs, Gr 5 | 0 | 0
  MCT Disorder AEs, Gr 1 (spell out) | 36 | 28
  MCT Disorder AEs, Gr 2 | 44 | 12
  MCT Disorder AEs, Gr 3 | 12 | 3
  MCT Disorder AEs, Gr 4 | 0 | 0
  MCT Disorder AEs, Gr 5 | 0 | 0
  GDASC AEs, Gr 1 (spell out) | 51 | 47
  GDASC AEs, Gr 2 | 28 | 23
  GDASC AEs, Gr 3 | 9 | 6
  GDASC AEs, Gr 4 | 0 | 0
  GDASC AEs, Gr 5 | 0 | 0
  Skin and Subcutaneous Tissue Disorder AEs, Gr 1 | 25 | 29
  Skin and Subcutaneous Tissue Disorder AEs, Gr 2 | 60 | 70
  Skin and Subcutaneous Tissue Disorder AEs, Gr 3 | 3 | 2
  Skin and Subcutaneous Tissue Disorder AEs, Gr 4 | 0 | 0
  Skin and Subcutaneous Tissue Disorder AEs, Gr 5 | 0 | 0
  Nervous System Disorder AEs, Gr 1 | 45 | 52
  Nervous System Disorder AEs, Gr 2 | 27 | 25
  Nervous System Disorder AEs, Gr 3 | 7 | 6
  Nervous System Disorder AEs, Gr 4 | 0 | 1
  Nervous System Disorder AEs, Gr 5 | 0 | 0
  Blood & Lymphatic System Disorder AEs, Gr 1 | 4 | 2
  Blood & Lymphatic System Disorder AEs, Gr 2 | 13 | 15
  Blood & Lymphatic System Disorder AEs, Gr 3 | 20 | 15
  Blood & Lymphatic System Disorder AEs, Gr 4 | 15 | 21
  Blood & Lymphatic System Disorder AEs, Gr 5 | 0 | 0
  Laboratory Investigation AEs, Gr 1 | 11 | 5
  Laboratory Investigation AEs, Gr 2 | 5 | 10
  Laboratory Investigation AEs, Gr 3 | 7 | 9
  Laboratory Investigation AEs, Gr 4 | 6 | 3
  Laboratory Investigation AEs, Gr 5 | 0 | 0
  Metabolism & Nutrition Disorder AEs, Gr 1 | 13 | 8
  Metabolism & Nutrition Disorder AEs, Gr 2 | 9 | 8
  Metabolism & Nutrition Disorder AEs, Gr 3 | 0 | 1
  Metabolism & Nutrition Disorder AEs, Gr 4 | 0 | 0
  Metabolism & Nutrition Disorder AEs, Gr 5 | 0 | 0
  RTM Disorder AEs, Gr 1 (spell out) | 18 | 17
  RTM Disorder AEs, Gr 2 | 1 | 6
  RTM Disorder AEs, Gr 3 | 1 | 1
  RTM Disorder AEs, Gr 4 | 1 | 3
  RTM Disorder AEs, Gr 5 | 0 | 0
  Infections & Infestations AEs, Gr 1 | 9 | 6
  Infections & Infestations AEs, Gr 2 | 8 | 7
  Infections & Infestations AEs, Gr 3 | 3 | 1
  Infections & Infestations AEs, Gr 4 | 0 | 1
  Infections & Infestations, Gr 5 | 0 | 0
  Psychiatric Disorder AEs, Gr 1 | 13 | 15
  Psychiatric Disorder AEs, Gr 2 | 3 | 2
  Psychiatric Disorder AEs, Gr 3 | 2 | 0
  Psychiatric Disorder AEs, Gr 4 | 0 | 0
  Psychiatric Disorder AEs, Gr 5 | 0 | 0
  Vascular Disorder AEs, Gr 1 | 12 | 17
  Vascular Disorder AEs, Gr 2 | 5 | 3
  Vascular Disorder AEs, Gr 3 | 1 | 0
  Vascular Disorder AEs, Gr 4 | 0 | 2
  Vascular Disorder AEs, Gr 5 | 0 | 0
  Eye Disorder AEs, Gr 1 | 14 | 10
  Eye Disorder AEs, Gr 2 | 1 | 1
  Eye Disorder AEs, Gr 3 | 0 | 0
  Eye Disorder AEs, Gr 4 | 0 | 0
  Eye Disorder AEs, Gr 5 | 0 | 0
  Immune System Disorder AEs, Gr 1 | 3 | 2
  Immune System Disorder AEs, Gr 2 | 2 | 0
  Immune System Disorder AEs, Gr 3 | 0 | 0
  Immune System Disorder AEs, Gr 4 | 2 | 0
  Immune System Disorder AEs, Gr 5 | 0 | 0
  Reproductive System and Breast Disorders, Gr 1 | 2 | 1
  Reproductive System and Breast Disorders, Gr 2 | 3 | 1
  Reproductive System and Breast Disorders, Gr 3 | 1 | 0
  Reproductive System and Breast Disorders, Gr 4 | 0 | 0
  Reproductive System and Breast Disorders, Gr 5 | 0 | 0
  Cardiac Disorder AEs, Gr 1 | 1 | 3
  Cardiac Disorder AEs, Gr 2 | 0 | 2
  Cardiac Disorder AEs, Gr 3 | 3 | 0
  Cardiac Disorder AEs, Gr 4 | 0 | 1
  Cardiac Disorder AEs, Gr 5 | 0 | 0
  Ear and Labyrinth Disorder AEs, Gr 1 | 1 | 4
  Ear and Labyrinth Disorder AEs, Gr 2 | 3 | 0
  Ear and Labyrinth Disorder AEs, Gr 3 | 0 | 0
  Ear and Labyrinth Disorder AEs, Gr 4 | 0 | 0
  Ear and Labyrinth Disorder AEs, Gr 5 | 0 | 0
  Renal and Urinary Disorder AEs, Gr 1 | 2 | 1
  Renal and Urinary Disorder AEs, Gr 2 | 0 | 0
  Renal and Urinary Disorder AEs, Gr 3 | 0 | 0
  Renal and Urinary Disorder AEs, Gr 4 | 0 | 0
  Renal and Urinary Disorder AEs, Gr 5 | 0 | 0
  Injury, Poisoning&Procedural Complication AEs,Gr 1 | 0 | 1
  Injury, Poisoning&Procedural Complication AEs,Gr 2 | 1 | 0
  Injury, Poisoning&Procedural Complication AEs,Gr 3 | 0 | 0
  Injury, Poisoning&Procedural Complication AEs,Gr 4 | 0 | 0
  Injury, Poisoning&Procedural Complication AEs,Gr 5 | 0 | 0
  Hepatobiliary Disorder AEs, Gr 1 | 0 | 0
  Hepatobiliary Disorder AEs, Gr 2 | 0 | 0
  Hepatobiliary Disorder AEs, Gr 3 | 0 | 0
  Hepatobiliary Disorder AEs, Gr 4 | 0 | 1
  Hepatobiliary Disorder AEs, Gr 5 | 0 | 0
  NBMUCP AEs, Gr 1 | 0 | 0
  NBMUCP AEs, Gr 2 | 0 | 1
  NBMUCP AEs, Gr 3 | 0 | 0
  NBMUCP AEs, Gr 4 | 0 | 0
  NBMUCP AEs, Gr 5 | 0 | 0

13. Secondary Outcome: On-Study Hematology: Worst Common Terminology Criteria of Adverse Events (CTCAE Version 3) Grade Per Participant in Ixabepilone/Paclitaxel Phase
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. Graded by National Cancer Institute Common Terminology Criteria for Adverse Events v3.0. (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death)
Time Frame: prior to the first study treatment, at the beginning of each subsequent cycle, weekly during the treatment period and a minimum of 4 weeks after the last dose of 12 weeks of study therapy during ixabepilone or paclitaxel treatment phase
Population: Ixabepilone/Paclitaxel treated participants for whom on-study labs were recorded.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 143 | 143
Participants
  White Blood Cells (WBC), Grade 0 | 32 | 32
  WBC, Grade 1 | 27 | 63
  WBC, Grade 2 | 32 | 41
  WBC, Grade 3 | 44 | 7
  WBC, Grade 4 | 8 | 0
  WBC, Grade 1-4 | 111 | 111
  WBC, Grade 3-4 | 52 | 7
  Absolute Neutrophil Count (ANC), Grade 0 | 33 | 66
  ANC, Grade 1 | 23 | 41
  ANC, Grade 2 | 28 | 24
  ANC, Grade 3 | 36 | 12
  ANC, Grade 4 | 23 | 0
  ANC, Grade 1-4 | 110 | 77
  ANC, Grade 3-4 | 59 | 12
  Platelets, Grade 0 | 109 | 134
  Platelets, Grade 1 | 33 | 6
  Platelets, Grade 2 | 0 | 2
  Platelets, Grade 3 | 1 | 1
  Platelets, Grade 4 | 0 | 0
  Platelets, Grade 1-4 | 34 | 9
  Platelets, Grade 3-4 | 1 | 1
  Hemoglobin, Grade 0 | 13 | 8
  Hemoglobin, Grade 1 | 77 | 91
  Hemoglobin, Grade 2 | 51 | 37
  Hemoglobin, Grade 3 | 2 | 6
  Hemoglobin, Grade 4 | 0 | 1
  Hemoglobin, Grade 1-4 | 130 | 135
  Hemoglobin, Grade 3-4 | 2 | 7

14. Primary Outcome: Percentage of Participants Achieving Pathologic Complete Response (pCR) in Biomarker-Defined Populations
Description: Beta III tubulin positivity determined by cross-validation method. Optimal cutoff: ≥46% tumor cells staining at 2 plus or 3 plus intensity (corresponding Beta III tubulin positivity=39.4%). Pre-specified cutoff of Beta III tubulin positivity: ≥50% 2plus or 3plus cells (corresponding prevalence=38.5%). Optimal cutoffs for TACC3 and CAPG positivity determined by cross-validation method: 6.889 and 6.844 [log2 normalized intensity units], respectively (corresponding to prevalence rates of 43.3% and 44.3%).
Time Frame: as for outcome 6
Population: For all subgroups other than Beta-III positive/negative subgroup based on a pre-determined cutoff, results were estimated using a cross-validation method (a resampling based technique, making individual sample size [N] not applicable).
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 148 | 147
Percentage of Participants
  Beta-III positive subgroup (cross-validation) | 35.9 [20.6 to 53.2] | 36.1 [23.3 to 56]
  Beta-III negative subgroup (cross-validation) | 17.4 [10.3 to 27.1] | 22.4 [13.1 to 32.0]
  Beta-III positive subgroup (n=43, 42) | 34.9 [22.9 to 48.5] | 35.7 [23.5 to 49.5]
  Beta-III negative subgroup (n=71, 75) | 18.3 [11.2 to 27.5] | 22.7 [15.0 to 32.0]
  TACC3 positive subgroup (cross-validation) | 30.1 [18.1 to 37.9] | 29.4 [19.6 to 47.2]
  TACC3 negative subgroup (cross-validation) | 19.8 [10.8 to 30.7] | 27.0 [13.2 to 41.4]
  CAPG positive subgroup (cross-validation) | 30.7 [18.9 to 47.4] | 35.3 [24.0 to 49.9]
  CAPG negative subgroup (cross-validation) | 20.4 [11.4 to 31.5] | 20.7 [9.1 to 44.3]

15. Secondary Outcome: On-Study Liver Function: Worst Common Terminology Criteria of Adverse Events (CTCAE Version 3) Grade Per Participant in Ixabepilone/Paclitaxel Phase
Description: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST). AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. Graded by National Cancer Institute Common Terminology Criteria for Adverse Events v3.0. (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death)
Time Frame: prior to the first study treatment, at the beginning of each subsequent cycle, weekly during the treatment period and a minimum of 4 weeks after the last dose of study therapy during ixabepilone or paclitaxel treatment phase
Population: Ixabepilone/Paclitaxel treated participants for whom on-study labs were recorded; n=number of participants with specific laboratory evaluation.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 143 | 143
Participants
  ALT, Grade 0 (n=142, 140) | 72 | 52
  ALT, Grade 1 (n=142, 140) | 54 | 59
  ALT, Grade 2 (n=142, 140) | 13 | 22
  ALT, Grade 3 (n=142, 140) | 3 | 7
  ALT, Grade 4 (n=142, 140) | 0 | 0
  ALT, Grade 1-4 (n=142, 140) | 70 | 88
  ALT, Grade 3-4 (n=142, 140) | 3 | 7
  AST, Grade 0 (n=141, 140) | 85 | 64
  AST, Grade 1 (n=141, 140) | 51 | 64
  AST, Grade 2 (n=141, 140) | 4 | 9
  AST, Grade 3 (n=141, 140) | 1 | 3
  AST, Grade 4 (n=141, 140) | 0 | 0
  AST, Grade 1-4 (n=141, 140) | 56 | 76
  AST, Grade 3-4 (n=141, 140) | 1 | 3
  Alkaline Phosphatase, Grade 0 (n=141, 140) | 114 | 117
  Alkaline Phosphatase, Grade 1 (n=141, 140) | 27 | 23
  Alkaline Phosphatase, Grade 2 (n=141, 140) | 0 | 0
  Alkaline Phosphatase, Grade 3 (n=141, 140) | 0 | 0
  Alkaline Phosphatase, Grade 4 (n=141, 140) | 0 | 0
  Alkaline Phosphatase, Grade 1-4 (n=141, 140) | 27 | 23
  Alkaline Phosphatase, Grade 3-4 (n=141, 140) | 0 | 0
  Total Bilirubin, Grade 0 (n=142, 140) | 137 | 131
  Total Bilirubin, Grade 1 (n=142, 140) | 4 | 8
  Total Bilirubin, Grade 2 (n=142, 140) | 0 | 0
  Total Bilirubin, Grade 3 (n=142, 140) | 1 | 0
  Total Bilirubin, Grade 4 (n=142, 140) | 0 | 1
  Total Bilirubin, Grade 1-4 (n=142, 140) | 5 | 9
  Total Bilirubin, Grade 3-4 (n=142, 140) | 1 | 1

16. Secondary Outcome: On-Study Renal Function: Worst Common Terminology Criteria of Adverse Events (CTCAE Version 3) Grade Per Participant in Ixabepilone/Paclitaxel Phase
Description: as for outcome 13
Time Frame: as for outcome 13
Population: Ixabepilone/Paclitaxel treated participants for whom on-study labs were recorded.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 142 | 139
Participants
  Creatinine, Grade 0 | 136 | 135
  Creatinine, Grade 1 | 6 | 3
  Creatinine, Grade 2 | 0 | 1
  Creatinine, Grade 3 | 0 | 0
  Creatinine, Grade 4 | 0 | 0
  Creatinine, Grade 1-4 | 6 | 4
  Creatinine, Grade 3-4 | 0 | 0

17. Secondary Outcome: Number of Participants by Dose for AC
Time Frame: 12 weeks (4 3-week cycles)
Population: ixabepilone- and paclitaxel-treated participants
Measure: Number; unit: participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 145 | 144
participants
  Dose 1 (Week 3) | 145 | 144
  Dose 2 (Week 6) | 145 | 144
  Dose 3 (Week 9) | 145 | 142
  Dose 4 (Week 12) | 143 | 141

18. Secondary Outcome: Number of Participants by Dose for Ixabepilone/Paclitaxel
Time Frame: 12 weeks (4 3-week cycles for ixabepilone and 12 weekly doses for paclitaxel)
Population: ixabepilone- and paclitaxel-treated participants
Measure: Number; unit: participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 145 | 144
participants
  Dose 1 (Week 3, ixabepilone; Week 1 paclitaxel) | 145 | 144
  Dose 2 (Week 6, ixabepilone; Week 2 paclitaxel) | 139 | 142
  Dose 3 (Week 9, ixabepilone; Week 3 paclitaxel) | 130 | 139
  Dose 4 (Week 12, ixabepilone; Week 4 paclitaxel) | 124 | 139
  Dose 5 (Week 5 paclitaxel) | 0 | 135
  Dose 6 (Week 6 paclitaxel) | 0 | 135
  Dose 7 (Week 7 paclitaxel) | 0 | 132
  Dose 8 (Week 8 paclitaxel) | 0 | 131
  Dose 9 (Week 9 paclitaxel) | 0 | 129
  Dose 10 (Week 10 paclitaxel) | 0 | 128
  Dose 11 (Week 11 paclitaxel) | 0 | 123
  Dose 12 (Week 12 paclitaxel) | 0 | 118

19. Secondary Outcome: Reason for First Dose Reduction of AC
Time Frame: 12 weeks (4 3-week cycles)
Population: ixabepilone- and paclitaxel-treated participants with at least 2 courses of AC
Measure: Number; unit: participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 145 | 144
participants
  Participants with at least 1 dose reduction of AC | 5 | 7
  Adverse Event | 1 | 3
  Hematologic Toxicity | 3 | 3
  Non-Hematologic Toxicity | 0 | 1
  Not Reported | 1 | 0

20. Secondary Outcome: Reason for First Dose Reduction of Ixabepilone/Paclitaxel
Time Frame: 12 weeks (4 3-week cycles for ixabepilone and 12 weekly doses for paclitaxel)
Population: ixabepilone- and paclitaxel-treated participants with at least 2 courses of Ixabepilone/Paclitaxel
Measure: Number; unit: participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 145 | 144
participants
  Participants with at least 1 dose reduction | 18 | 18
  Adverse Event | 10 | 3
  Hematologic Toxicity | 2 | 0
  Non-Hematologic Toxicity | 0 | 4
  Not Reported | 1 | 2
  Peripheral Neuropathy | 5 | 9

21. Secondary Outcome: Number of Participants With Course Delay and Reason for Delay for AC
Time Frame: 12 weeks (4 3-week cycles)
Population: ixabepilone- and paclitaxel-treated participants with at least 2 courses of AC
Measure: Number; unit: participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 145 | 144
participants
  Participants with at least 1 dose delay | 41 | 43
  Administrative Reason | 5 | 6
  Adverse Event | 6 | 10
  Hematologic Toxicity | 17 | 10
  Non-Hematologic Toxicity | 3 | 2
  Not Reported | 14 | 16
  Other | 3 | 1
  Subject Request | 2 | 0

22. Secondary Outcome: Number of Participants With Dose Delay and Reason for Dose Delay for Ixabepilone/Paclitaxel
Time Frame: 12 weeks (4 3-week cycles for ixabepilone and 12 weekly doses for paclitaxel)
Population: ixabepilone- and paclitaxel-treated participants with at least 2 courses of Ixabepilone/Paclitaxel
Measure: Number; unit: participants
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 145 | 144
participants
  Participants with at least 1 dose delay | 31 | 51
  Administrative Reason | 3 | 5
  Adverse Event | 6 | 15
  Hematologic Toxicity | 10 | 15
  Non-Hematologic Toxicity | 0 | 7
  Not Reported | 13 | 8
  Other | 3 | 8
  Peripheral Neuropathy | 0 | 1
  Subject Request | 0 | 3

23. Primary Outcome: Percentage of Participants Achieving Pathologic Complete Response (pCR) in 20- and 26-Gene Model Subgroups
Description: For each of the 2 biomarker sets (20-gene or 26-gene), a multi-gene model was built using penalized logistic regression on all pharmacogenomic evaluable subjects for each treatment arm separately. Receiver Operating Characteristic (ROC) plots for separate arm using 5 fold cross validation were generated. ROC for separate arms using cross over were also added. Further analysis on the multiple gene models (as mentioned in the SAP) was planned only based on the initial findings from the 2 ROC plots. For 20- and 26-gene models, ROC curves generated for each study arm did not indicate that these multi-gene models differentially predicted for pCR between the treatment arms, so further analyses to estimate the optimal cut-off and the pCR rates were not conducted.
Time Frame: as for outcome 6
Population: For 20- and 26-gene models, ROC curves generated for each study arm did not indicate that these multi-gene models differentially predicted for pCR between the treatment arms, so further analyses to estimate the optimal cut-off and the pCR rates were not conducted.
Arm/Group | Ixabepilone | Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events are reported for randomized population.
Arm/Group | Ixabepilone | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 17/145 | 11/144
Other Adverse Events (participants affected / at risk) | 128/145 | 117/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=145) | Paclitaxel (N=144)
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
CRANIAL NEUROPATHY (Nervous system disorders) | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
CEREBRAL VENOUS THROMBOSIS (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
GALLSTONE ILEUS (Gastrointestinal disorders) | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 3 | 0
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 3
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1
NON-CARDIOGENIC PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
FATIGUE (General disorders) | 2 | 1
PYREXIA (General disorders) | 0 | 3
SUDDEN DEATH (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=145) | Paclitaxel (N=144)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 | 12
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 9
HOT FLUSH (Vascular disorders) | 8 | 12
INSOMNIA (Psychiatric disorders) | 16 | 17
HEADACHE (Nervous system disorders) | 6 | 9
DYSGEUSIA (Nervous system disorders) | 2 | 8
PARAESTHESIA (Nervous system disorders) | 10 | 4
NEUROPATHY PERIPHERAL (Nervous system disorders) | 24 | 23
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 27 | 44
NAUSEA (Gastrointestinal disorders) | 27 | 18
VOMITING (Gastrointestinal disorders) | 14 | 5
DIARRHOEA (Gastrointestinal disorders) | 24 | 19
STOMATITIS (Gastrointestinal disorders) | 6 | 11
CONSTIPATION (Gastrointestinal disorders) | 9 | 9
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 | 9
NEUTROPENIA (Blood and lymphatic system disorders) | 28 | 15
RASH (Skin and subcutaneous tissue disorders) | 13 | 16
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 9
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 7 | 12
MYALGIA (Musculoskeletal and connective tissue disorders) | 43 | 18
BONE PAIN (Musculoskeletal and connective tissue disorders) | 30 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 34 | 15
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 7
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 16 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 19
PAIN (General disorders) | 10 | 8
FATIGUE (General disorders) | 27 | 24
PYREXIA (General disorders) | 6 | 10
ASTHENIA (General disorders) | 13 | 10
MUCOSAL INFLAMMATION (General disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.